CLINICAL TRIAL: NCT07231926
Title: The Effects of Intrathecal Morphine in Addition to Serratus Anterior Plane Block and Dexmedetomidine on Postoperative Recovery (QoR-15) and Systemic Inflammation in Video-Assisted Thoracoscopic Surgery: A Randomized Controlled Trial
Brief Title: Intrathecal Morphine for Recovery and Outcomes After VATS
Acronym: IMPROVE-VATS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, irem ateş, Principal Investigator İrem Ateş, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/614; 2025/2 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-09-19; First posted 2025-11-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain Management in Video-Assisted Thoracoscopic Surgery
Keywords: Video-Assisted Thoracoscopic Surgery; Postoperative Analgesia; Intrathecal Morphine; Patient-Controlled Analgesia (PCA); Thoracic Surgery Pain Management
MeSH Terms: interventions — Saposins; Population Groups; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups in a 1:1 ratio: Group ITM + SAPB + Dexmedetomidine and Group SAPB + Dexmedetomidine.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and postoperative data collectors will be blinded to group allocation. The anesthesiologist performing the intervention will be aware of the allocation due to the nature of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ITM + SAPB + Dex (Experimental): Before induction, 200 µg intrathecal morphine via a 27G Sprotte spinal needle from L3-L4; intraoperative 1 g paracetamol IV and 50 mg dexketoprofen IV; dexmedetomidine 0.5 µg/kg loading (15 min) followed by a 0.5 µg/kg/h infusion; unilateral SAPB with 30 mL of 0.25% bupivacaine under ultrasound guidance at the end of surgery; basal tramadol PCA without infusion IV in the PACU (20 mg each bolus, maximum 200 mg/24 h); if necessary, 50 mg tramadol IV for VAS>4.
  Interventions: Drug: Intrathecal Morphine; Procedure: Serratus Anterior Plane Block (SAPB) group; Drug: Dexmedetomidine
- SAPB + Dex (No ITM) (Active Comparator): Same protocol, but no intrathecal morphine. Intraoperatively, 1 g paracetamol IV and 50 mg dexketoprofen IV; dexmedetomidine 0.5 µg/kg loading dose (15 min) followed by a 0.5 µg/kg/h infusion; unilateral SAPB with 30 mL of 0.25% bupivacaine at the end of surgery; basal intravenous tramadol PCA (20 mg each bolus, maximum 200 mg/24 h) in the PACU; if necessary, 50 mg tramadol IV for VAS >4.
  Interventions: Procedure: Serratus Anterior Plane Block (SAPB) group; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Intrathecal Morphine — 200 µg morphine sulfate, single-dose via L3-L4, 27G Sprotte spinal needle, prior to induction.
  Arms: ITM + SAPB + Dex
Procedure: Serratus Anterior Plane Block (SAPB) group — Ultrasound-guided unilateral SAPB at end of surgery with 30 mL 0.25% bupivacaine.
Drug: Dexmedetomidine — Loading dose 0.5 µg/kg over 15 minutes, then 0.5 µg/kg/h continuous infusion intraoperatively.

SUMMARY:
This study will compare two different methods of pain management in patients undergoing video-assisted thoracoscopic surgery (VATS). One group will receive a combination of spinal morphine, nerve block, and dexmedetomidine, while the other group will receive a nerve block and dexmedetomidine without spinal morphine. All patients will receive standard pain medications after surgery. The purpose is to see if adding spinal morphine improves pain control and recovery after surgery.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, double-blind clinical trial evaluating the efficacy of intrathecal morphine in combination with serratus anterior plane block (SAPB) and dexmedetomidine infusion for postoperative analgesia in patients undergoing elective video-assisted thoracoscopic surgery (VATS). Eligible patients are ASA I-II, aged 18-70 years, with BMI < 35 kg/m². Patients will be randomized into two groups using a computer-generated sequence. The intervention group will receive intrathecal morphine (200 µg) in addition to SAPB and dexmedetomidine, while the control group will receive SAPB and dexmedetomidine alone. The primary outcome is postoperative pain scores (VAS) within the first 24 hours. Secondary outcomes include opioid consumption, quality of recovery, and incidence of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Elective video-assisted thoracoscopic surgery (VATS) planned
* Age 18-70 years
* ASA physical status I-III
* Body mass index (BMI) <35 kg/m²

Exclusion Criteria:

* Coagulopathy
* Opioid dependence or intolerance
* Allergy to local anesthetics
* Contraindications to neuraxial blockade
* Chronic pain history
* Renal or hepatic failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-15 (QoR-15) Score | Measured 24 hours after surgery
  The Quality of Recovery-15 (QoR-15) questionnaire is a validated 15-item instrument that assesses patient-centered postoperative recovery, including pain, physical comfort, emotional state, and overall wellbeing. The total score ranges from 0 to 150, with higher scores indicating better recovery.

SECONDARY OUTCOMES:
Time to First Rescue Opioid | Within 24 hours postoperatively
  Duration (in hours) from the end of surgery to the first administration of rescue opioid (intravenous tramadol) when the Visual Analog Scale (VAS) pain score exceeds 4.
Postoperative Pain Scores (VAS) | From postoperative hour 2 to hour 24.
  Postoperative pain intensity will be evaluated using the Visual Analog Scale (VAS), a 10-cm line ranging from 0 (no pain) to 10 (worst imaginable pain). Both active (movement) and passive (rest) VAS scores will be recorded at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, and 24 hours after surgery. Higher scores indicate more severe pain.
Total Opioid Consumption | 24 hours postoperatively
  Cumulative opioid consumption (including PCA tramadol, subcutaneous morphine, and rescue IV tramadol) within 24 hours postoperatively, reported in mg.
Intraoperative Complications | During surgery
  Occurrence of bradycardia, hypotension, or other anesthesia-related intraoperative adverse events.
Postoperative Adverse Effects | 24 hours postoperatively
  Incidence of nausea, vomiting, pruritus, respiratory depression, or other opioid-related side effects during the first 24 hours postoperatively.
Serum Interleukin-6 (IL-6) Level | Preoperatively and at 24 hours postoperatively
  Serum IL-6 levels (pg/mL) will be measured to evaluate the systemic inflammatory response associated with surgical stress.
Neutrophil-to-Lymphocyte Ratio (NLR) | Preoperatively and at 24 hours postoperatively
  The neutrophil-to-lymphocyte ratio (NLR) will be calculated to evaluate postoperative inflammatory status and its correlation with pain intensity and functional recovery.
Serum C-reactive Protein (CRP) Level | Preoperatively and at 24 hours postoperatively.
  Serum CRP levels (mg/L) will be measured to assess postoperative systemic inflammation.
Platelet-to-Lymphocyte Ratio (PLR) | Preoperatively and at 24 hours postoperatively.
  The platelet-to-lymphocyte ratio (PLR) will be calculated as a marker of postoperative inflammation and its correlation with pain level and recovery quality.
Lymphocyte-to-Monocyte Ratio (LMR) | Preoperatively and at 24 hours postoperatively.
  The lymphocyte-to-monocyte ratio (LMR) will be calculated to assess systemic immune response in relation to postoperative recovery.
Systemic Immune-Inflammation Index (SII) | Preoperatively and at 24 hours postoperatively.
  The systemic immune-inflammation index (SII) will be calculated as platelet × neutrophil / lymphocyte, providing an integrated indicator of postoperative inflammatory and immune status.

CONTACTS AND LOCATIONS:
Overall Officials: İREM ATEŞ, Principal Investigator — Ataturk University; Nuray Uzun, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study involves sensitive patient health information, and data confidentiality will be strictly maintained according to institutional ethical guidelines.

REFERENCES:
- [Background] Jiao Y, Zhang X, Liu M, Sun Y, Ma Z, Gu X, Gu W, Zhu W. Systemic immune-inflammation index within the first postoperative hour as a predictor of severe postoperative complications in upper abdominal surgery: a retrospective single-center study. BMC Gastroenterol. 2022 Aug 27;22(1):403. doi: 10.1186/s12876-022-02482-9. PMID 36030214
- [Background] Xu N, Zhang JX, Zhang JJ, Huang Z, Mao LC, Zhang ZY, Jin WD. The prognostic value of the neutrophil-to-lymphocyte ratio (NLR) and platelet-to-lymphocyte ratio (PLR) in colorectal cancer and colorectal anastomotic leakage patients: a retrospective study. BMC Surg. 2025 Feb 5;25(1):57. doi: 10.1186/s12893-024-02708-5. PMID 39910526
- [Background] Rettig TC, Verwijmeren L, Dijkstra IM, Boerma D, van de Garde EM, Noordzij PG. Postoperative Interleukin-6 Level and Early Detection of Complications After Elective Major Abdominal Surgery. Ann Surg. 2016 Jun;263(6):1207-12. doi: 10.1097/SLA.0000000000001342. PMID 26135695
- [Background] Huang ZY, Huang Q, Wang LY, Lei YT, Xu H, Shen B, Pei FX. Normal trajectory of Interleukin-6 and C-reactive protein in the perioperative period of total knee arthroplasty under an enhanced recovery after surgery scenario. BMC Musculoskelet Disord. 2020 Apr 21;21(1):264. doi: 10.1186/s12891-020-03283-5. PMID 32316949
- [Background] Yoon SH, Bae J, Yoon S, Na KJ, Lee HJ. Correlation Between Pain Intensity and Quality of Recovery After Video-Assisted Thoracic Surgery for Lung Cancer Resection. J Pain Res. 2023 Oct 2;16:3343-3352. doi: 10.2147/JPR.S426570. eCollection 2023. PMID 37808464
- [Background] Mugabure Bujedo B. A clinical approach to neuraxial morphine for the treatment of postoperative pain. Pain Res Treat. 2012;2012:612145. doi: 10.1155/2012/612145. Epub 2012 Jul 2. PMID 23002426
- [Background] Sibanyoni M, Biyase N, Motshabi Chakane P. The use of intrathecal morphine for acute postoperative pain in lower limb arthroplasty surgery: a survey of practice at an academic hospital. J Orthop Surg Res. 2022 Jun 21;17(1):323. doi: 10.1186/s13018-022-03215-0. PMID 35729586
- [Background] Meng G, Chen W, Shi D, Mei B, Liu X. Superficial vs. deep serratus anterior plane block for analgesia in patients undergoing single-port video-assisted thoracoscopic surgery: A randomized prospective trial. J Clin Anesth. 2025 Sep;106:111950. doi: 10.1016/j.jclinane.2025.111950. Epub 2025 Jul 31. PMID 40749388
- [Background] Liu Y, Liang F, Liu X, Shao X, Jiang N, Gan X. Dexmedetomidine Reduces Perioperative Opioid Consumption and Postoperative Pain Intensity in Neurosurgery: A Meta-analysis. J Neurosurg Anesthesiol. 2018 Apr;30(2):146-155. doi: 10.1097/ANA.0000000000000403. PMID 28079737
- [Background] Liu Y, Zhao G, Zang X, Lu F, Liu P, Chen W. Effect of dexmedetomidine on opioid consumption and pain control after laparoscopic cholecystectomy: a meta-analysis of randomized controlled trials. Wideochir Inne Tech Maloinwazyjne. 2021 Sep;16(3):491-500. doi: 10.5114/wiitm.2021.104197. Epub 2021 Mar 8. PMID 34691300